CLINICAL TRIAL: NCT00810433
Title: A Clinical Safety and Feasibility Study of the GO-LIF® Approach
Brief Title: A Clinical Study of the GO-LIF® Approach for Lumbar Spinal Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mazor Robotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-102; NCT00786955 (obsolete NCT alias)
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Procedure: GO-LIF - Guided Oblique Lumbar Interbody Fusion

INTERVENTIONS:
Procedure: GO-LIF - Guided Oblique Lumbar Interbody Fusion — All patients will undergo single-level instrumented interbody spinal fusion surgery with instrumentation.
  Upon induction of general anesthesia, the patient will be positioned prone on a radiolucent operating table and prepared according to standard hospital procedure. An interbody fusion will be performed according to standard procedure and as indicated by the surgeon. The interbody fusion portion of the surgery will be carried out using any current technique - such as PLIF, TLIF, PLF, PLLF, XLIF or ALIF. The fusion strategy can be performed in an open or minimally invasive manner, as indicated. The interbody device will be inserted after the screws trajectory will be drilled and a 4.5mm Trajectory holder is in place. This will assure the surgeon that no collision will occur between the interbody and the screws.
  Upon completion of the fusion stage of the surgery, SpineAssist will be used to introduce the GO-LIF screws for fixation of the spinal levels to be fused.
  Other Names: Mazor; SpineAssist; GO-LIF

SUMMARY:
The purpose of this study is to collect data regarding the safety and feasibility of the GO-LIF procedure for spinal fixation and stabilization, in conjunction with conventional approaches for interbody lumbar fusion. This is in order to allow for evidence-based comparison to pedicle-screw-based techniques as described in the literature.

ELIGIBILITY:
Inclusion Criteria

1. Men and women, 18-80 years of age.
2. The capability to comprehend the nature and rationale of the study and to consent to participating in the study.
3. Unequivocal medical indication for the fixation surgery of a single motion segment of the lumbar spine.
4. Correct coronal profile of the lumbar spine. An asymmetric collapse of the disk space in the coronal plane between the vertebral bodies envisioned for instrumentation is by itself not an exclusion criterion.

Or any of criteria below:

1. Patients with Grade II or Grade III spondylolisthesis in the sagittal plane with preserved or normal sagittal alignment requiring single-level instrumented interbody fusion from L1 to S1. (Not excluding patient with a need to decompression)
2. Patients must have normal alignment of the spine in the coronal view. 2. The interbody fusion approach may be TLIF or PLIF or ALIF or other, as clinically indicated.

   3. The procedure may be combined with a Micro-decompression and/or Micro-discectomy and/or direct or indirect decompression and/or laminectomy or laminotomy and/or other procedures, as clinically indicated - as long as such procedures do not compromise the structural integrity of the pedicles of the inferior vertebra or the vertebral body of either vertebra of the levels involved..

   4. Patient is 18 years or more 5. Patient is willing and able to comply with study requirements

   Exclusion Criteria:
   1. Lumbar hyperlordosis > 70° between the end plate of the lumbar vertebral body 1 and the end plate of the sacral vertebral body 1.
   2. Deformities of the vertebral bodies envisioned for instrumentation or the sacrum.
   3. Spondylolisthesis > grade 2 acc. to Meyerding.
   4. Scoliosis and other deformities in the coronal plane.
   5. Fractures of the vertebrae envisioned for instrumentation.
   6. Osteoporosis or osteopenia (see below for examination criteria).
   7. Therapy with systemic corticosteroids or immunosuppressants.
   8. Bone metabolism diseases, such as osteomalacia or Paget's disease.
   9. Post inflammatory instability of the vertebral spine.
   10. State after radiation therapy of the relevant vertebral spine region.
   11. Current Marcoumar or heparin therapy for more than 6 months at the time of operation.
   12. Malignant diseases with or without bone metastases.
   13. Immunologic-inflammatory diseases (e.g., rheumatoid arthritis).
   14. Diabetes mellitus.
   15. Infectious diseases.
   16. BMI > 30.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The number, severity and causality of intra-operative and post-operative complications, with particular attention to nerve root irritation or injury. | prior to discharge from hospital
Number of significant cortical breaches (>4mm), as evidenced by visual examination of a post-operative CT scan. | Preferably prior to discharge from hospital, and no later than 1 month post-op
The number of procedures that were not completed, and the reasons and causality for non-completions. | Immediately post-op.

SECONDARY OUTCOMES:
Plain AP, Lateral and flexion-extension radiographs. The radiographs will be examined for: • Evidence of bridging trabecular bone between the involved motion segments • Translational motion <3mm; and •Angular motion <5 degrees. | 3, 6 and 12 months post-op.
Healthcare Outcomes: the visual analogue pain scale (VAS), the Oswestry disability index (ODI) and Swiss Spinal Stenosis (SSS) Questionnaire. | pre-op; 3, 6 and 12 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Isador H Lieberman, MD, MBA, FRCSC, Study Director — Texas Back Institute
Locations (10):
- Germany (8):
  - Dep. Of Neurosurgery , Charité-Universitätsmedizin Berlin, Campus Benjamin Franklin (CBF), Berlin
  - Dep. Of Orthopedic Helios Rosmann Klinik, Breisach
  - Dept. of Neurosurgery, Neurochirurgische Klinik Göttingen, Göttingen
  - Dept. of Neurosurgery, Klinikum Nordstadt Hannover, Hanover
  - Dep. Of Neurosurgery Universitaetsklinikum Mannheim, Mannheim
  - Krankenhaus Munchen Schwabing, Munich
  - Dep. Of Orthopedic Klinikum Grosshadern- LMU, Munich
  - Dep. Of Neurosurgery Paracelsus kliniken, Munich
- Israel (2):
  - Dept. of Orthopedics, Carmel Medical Center, Haifa
  - Dept. of Orthopedics Hadassah Medical Center - The Hebrew University, Jerusalem

REFERENCES:
- [Derived] Birkenmaier C, Suess O, Pfeiffer M, Burger R, Schmieder K, Wegener B. The European multicenter trial on the safety and efficacy of guided oblique lumbar interbody fusion (GO-LIF). BMC Musculoskelet Disord. 2010 Sep 6;11:199. doi: 10.1186/1471-2474-11-199. PMID 20819219